CLINICAL TRIAL: NCT02266381
Title: A Prospective and Randomized Comparison of Fluoroscopic, Sonographic or Combined Approach for Renal Access in Percutaneous Nephrolithotomy
Brief Title: A Prospective Comparison of Fluoroscopic, Sonographic or Combined Approach for Renal Access in Percutaneous Nephrolithotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Guohua Zeng, Vice President of the Hospital, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MRER(29)2014
Record Dates: First submitted 2014-10-13; First posted 2014-10-17 (Estimated); Results first posted 2016-11-09 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-09

CONDITIONS: Urolithiasis
Keywords: PCNL; MPCNL; guidance; puncture
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- US-guided group (Other): Patients in US-guided group undergo MPCNL using only US-guided renal access.
  Interventions: Procedure: US-guided renal access
- Fluoroscopy-guided group (Other): Patients in Fluoroscopy-guided group undergo MPCNL using only fluoroscopy-guided renal access.
  Interventions: Procedure: Fluoroscopy-guided renal access
- Combined-guided group (Other): Patients in Combined-guided group undergo MPCNL using US combined with fluoroscopy-guided renal access.
  Interventions: Procedure: US combined with fluoroscopy-guided renal access

INTERVENTIONS:
Procedure: US-guided renal access — Patients undergo MPCNL using only US-guided renal access.
  Arms: US-guided group
Procedure: Fluoroscopy-guided renal access — Patients undergo MPCNL using only fluoroscopy-guided renal access.
  Arms: Fluoroscopy-guided group
Procedure: US combined with fluoroscopy-guided renal access — Patients undergo MPCNL using US combined with fluoroscopy-guided renal access
  Arms: Combined-guided group

SUMMARY:
Purpose:

The aim of this present study is to compare the result of fluoroscopy, ultrasonography (US) and US combined with fluoroscopy in the guidance of minimally invasive percutaneous nephrolithotomy (MPCNL).

Methods:

The investigators will enroll 450 patients who are candidates for MPCNL in our study. By simple random sampling technique, patients will be assigned to three 150-patient groups (group 1, US-guided MPCNL, group 2, fluoroscopy-guided MPCNL and group 3, US combined with fluoroscopy-guided MPCNL). In addition to approaches in guidance of MPCNL, the rest of the procedure is the same in all three groups.The end point of the study is the comparison of outcome of procedure including stone free rate, transfusion rate, operation time, access time, length of stay and complications.

DETAILED DESCRIPTION:
Purpose:

Recently, PCNL or MPCNL is widely used as the most popular choice to treat patients with all types of renal stones. Successful puncture to the desired renal calyx is the key step for the operation. Nowadays puncture for renal access can be achieve using not only US guidance but fluoroscopy guidance as well. However, it is clear that there is a lack of randomized controlled data comparing fluoroscopy, US and US combined with fluoroscopy in the guidance of MPCNL. Consequently, we performed this randomized controlled trial to obtain higher grade evidence.The aim of this present study is to compare the result of fluoroscopy, US and US combined with fluoroscopy in the guidance of MPCNL.

Methods:

We will enroll 450 patients who are candidates for MPCNL in our study. By simple random sampling technique, patients will be assigned to three 150-patient groups (group 1, US-guided MPCNL, group 2, fluoroscopy-guided MPCNL and group 3, US combined with fluoroscopy-guided MPCNL).

All the patients will be diagnosed definitely before operations with kidney, ureter, and bladder (KUB), intravenous pyelography (IVP), US and/or CT.

All procedures are performed by urologists in our center, with assistance from an endourology fellow.

Surgical technique:

Under general or epidural anaesthesia, each patient is initially placed in the lithotomy position, and a 5 Fr ureteric catheter is advanced to the kidney and fixed with a 16 Fr Foley catheter. Then the patient is turned to the prone position.

Group 1: US-guided MPCNL The puncture is made with an 18-gauge needle using an ultrasound probe. After the desirable calix is reached, a flexible-tip guidewire is introduced. We attempt to manipulate the guidewire down to the ureter. If this is not successful, the second choice is to allow the guidewire to coil in a more distant calix. The length of the needle from skin to the collecting system is measured to ensure that the length of dilator is appropriate. The access tract is dilated from 8 Fr to a maximum 18/20 Fr using fascial dilator. We defined access to the collecting system as gaining entry to the targeted urinary system and desired calix.

Lithotripsy is performed using either pneumatic lithotriptor or holmium laser. When multiple nephrostomy tracts are necessary to remove the stones, same technique is employed for each of the tracts.

Complete stone clearance is confirmed using US at completion of the procedure. We routinely put a double J ureteral catheter into the ureter which is to be removed about 3-4 weeks later after the operation in the out-patients clinic. At the end of the procedure nephrostomy tubes are placed in both groups. The tubes are removed when the drainage from nephrostomy tubes being grossly clear.

Group 2 fluoroscopy-guided MPCNL Patients in group 2 have the standard fluoroscopy-guided renal access before MPCNL. Air or contrast medium is injected through the ureteral catheter, the target calix is identified. For tract dilatation fascial dilators are used under fluoroscopic guidance.

Complete stone clearance is confirmed fluoroscopically at completion of the procedure.

The rest of the procedure is the same as described for patients in group 1.

Group 3 US combined with fluoroscopy-guided MPCNL:

Under the guidance of ultrasound, the coaxial needle is placed in the desired calyx. A floppy-tipped guidewire is then passed through the needle into the collecting system. The working channel is then dilated under X-ray.

US and X-ray check for residual stone fragments are performed at the end of the procedure.

The rest of the procedure is the same as described for patients in group 1.

Data collection:

Data for the three groups -demographic characteristics, access success, access time, duration of radiation exposure, site of target calix, site of access, Hb decrease, duration of postoperative hospital stay, complications (modified Clavien system), stone clearance (SFR after single procedure and final SFR) and the need for auxiliary treatment - are compared.

The primary end point of the study is the comparison of outcome of procedure including stone free rate, transfusion rate, operation time, access time, length of stay and complications.

ELIGIBILITY:
Inclusion Criteria:

* Normal renal function.
* American society of Anesthesiology (ASA) score 1 and 2.
* Absence of congenital abnormalities.
* Kidney stones of diameter > 2.0cm (including multiple and staghorn stones)

Exclusion Criteria:

* Patients with congenital anomalies, e.g. ectopic kidney, polycystic, horseshoe, or malrotated kidney.
* Patients who underwent transplant or urinary diversion.
* Patients with solitary kidney.
* Patients will be excluded from the study if they undergoing MPCNL have purulent fluid in the initial puncture.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guohua Zeng, PH.D and M.D, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Department of Urology, Minimally Invasive Surgery Center, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Lu MH, Pu XY, Gao X, Zhou XF, Qiu JG, Si-Tu J. A comparative study of clinical value of single B-mode ultrasound guidance and B-mode combined with color doppler ultrasound guidance in mini-invasive percutaneous nephrolithotomy to decrease hemorrhagic complications. Urology. 2010 Oct;76(4):815-20. doi: 10.1016/j.urology.2009.08.091. Epub 2010 Jun 25. PMID 20579695
- [Background] Mozer P, Conort P, Leroy A, Baumann M, Payan Y, Troccaz J, Chartier-Kastler E, Richard F. Aid to percutaneous renal access by virtual projection of the ultrasound puncture tract onto fluoroscopic images. J Endourol. 2007 May;21(5):460-5. doi: 10.1089/end.2006.0168. PMID 17523896
- [Background] Yan S, Xiang F, Yongsheng S. Percutaneous nephrolithotomy guided solely by ultrasonography: a 5-year study of >700 cases. BJU Int. 2013 Nov;112(7):965-71. doi: 10.1111/bju.12248. Epub 2013 Jul 26. PMID 23889729
- [Background] Li X, Long Q, Chen X, He D, He H. Real-time ultrasound-guided PCNL using a novel SonixGPS needle tracking system. Urolithiasis. 2014 Aug;42(4):341-6. doi: 10.1007/s00240-014-0671-2. Epub 2014 Jun 26. PMID 24965272
- [Background] Agarwal M, Agrawal MS, Jaiswal A, Kumar D, Yadav H, Lavania P. Safety and efficacy of ultrasonography as an adjunct to fluoroscopy for renal access in percutaneous nephrolithotomy (PCNL). BJU Int. 2011 Oct;108(8):1346-9. doi: 10.1111/j.1464-410X.2010.10002.x. Epub 2011 Jan 20. PMID 21251187
- [Background] Opondo D, Gravas S, Joyce A, Pearle M, Matsuda T, Sun YH, Assimos D, Denstedt J, de la Rosette J. Standardization of patient outcomes reporting in percutaneous nephrolithotomy. J Endourol. 2014 Jul;28(7):767-74. doi: 10.1089/end.2014.0057. Epub 2014 Apr 16. PMID 24571713
- [Background] Basiri A, Ziaee AM, Kianian HR, Mehrabi S, Karami H, Moghaddam SM. Ultrasonographic versus fluoroscopic access for percutaneous nephrolithotomy: a randomized clinical trial. J Endourol. 2008 Feb;22(2):281-4. doi: 10.1089/end.2007.0141. PMID 18294034
- [Background] Desai M, Jain P, Ganpule A, Sabnis R, Patel S, Shrivastav P. Developments in technique and technology: the effect on the results of percutaneous nephrolithotomy for staghorn calculi. BJU Int. 2009 Aug;104(4):542-8; discussion 548. doi: 10.1111/j.1464-410X.2009.08472.x. Epub 2009 Mar 6. PMID 19298409
- [Derived] Zhu W, Li J, Yuan J, Liu Y, Wan SP, Liu G, Chen W, Wu W, Luo J, Zhong D, Qi D, Lei M, Zhong W, Zhang Z, He Z, Zhao Z, Lu S, Wu Y, Zeng G. A prospective and randomised trial comparing fluoroscopic, total ultrasonographic, and combined guidance for renal access in mini-percutaneous nephrolithotomy. BJU Int. 2017 Apr;119(4):612-618. doi: 10.1111/bju.13703. Epub 2016 Nov 28. PMID 27862806

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A prospective and randomized study was performed with patient enrollment from July 2014 to May 2015 in the First Affilated Hospital of Guangzhou Medical University. 450 patients were then randomized into three groups. 12 patients had purulent fluid in the kidney at initial punctures. These 12 patients were excluded from the analysis.
Pre-assignment Details: 549 consecutive patients were assessed for eligibility, 99 were excluded for not meeting the inclusion criteria.
Period: Overall Study
Arm/Group | US-guided Group | Fluoroscopy-guided Group | Combined-guided Group
Started | 150 | 150 | 150
Completed | 147 | 145 | 146
Not Completed | 3 | 5 | 4
Not completed — Physician Decision | 3 | 5 | 4

BASELINE CHARACTERISTICS:
Population: 450 patients were then randomized into three groups.12 patients had purulent fluid in the kidney at initial punctures. A nephrostomy tube was placed and MPCNL postponed to avoid septic complications. These 12 patients were excluded from the analysis. Finally, 438 patients were accrued in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | US-guided Group | Fluoroscopy-guided Group | Combined-guided Group | Total
Number analyzed (Participants) | 147 | 145 | 146 | 438
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (10.9) | 49.6 (11.3) | 48.8 (11.3) | 49.4 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 68 | 58 | 187
  Male | 86 | 77 | 88 | 251
Region of Enrollment [Number; unit: participants]
  China | 147 | 145 | 146 | 438

OUTCOME MEASURES:

1. Primary Outcome: Stone Free Rate
Description: Stone-free status is assessed by kidneys-ureter-bladder (KUB) or/ and noncontrast CT at day 1 after MPCNL. A stone-free state is defined as no residual stones of diameter >4 mm.
Time Frame: one day after MPCNL
Measure: Number; unit: Participants
Arm/Group | US-guided Group | Fluoroscopy-guided Group | Combined-guided Group
Number analyzed (Participants) | 147 | 145 | 146
Participants | 81 | 91 | 98

2. Secondary Outcome: Perioperative Complications
Description: Complication is defined as any adverse event occurred intraoperatively or ≤ 30 days postoperatively. Complications included fever, systemic Inflammatory Response Syndrome, septic shock, extravasations, bleeding necessitating transfusion, and sever bleeding necessitating selective renal artery embolization.
Time Frame: intraoperatively or ≤ 30 days postoperatively
Measure: Number; unit: Participants
Groups:
- US-guided Group: Patients in US-guided undergo MPCNL using only US-guided renal access.
- Combined Group: Patients in Combined group undergo MPCNL using US combined with fluoroscopy-guided renal access.
Arm/Group | US-guided Group | Fluoroscopy-guided Group | Combined Group
Number analyzed (Participants) | 147 | 145 | 146
Participants | 17 | 31 | 20

3. Secondary Outcome: Operation Time
Description: Operation time is defined as the time from puncture to the placement of the nephrostomy tube.
Time Frame: intraoperatively
Measure: Mean (Standard Deviation); unit: min
Arm/Group | US-guided Group | Fluoroscopy-guided Group | Combined-guided Group
Number analyzed (Participants) | 147 | 145 | 146
min | 60.6 (32.9) | 63.6 (32.5) | 66.3 (34.7)

4. Secondary Outcome: Change in Hemoglobin Concentration
Description: Change in hemoglobin concentration is assessed by comparing the preoperative hemoglobin level with 24-hour postoperative hemoglobin level.
Time Frame: within 24 hours after MPCNL
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | US-guided Group | Fluoroscopy-guided Group | Combined-guided Group
Number analyzed (Participants) | 147 | 145 | 146
g/L | 12.9 (16.0) | 14.5 (10.0) | 13.1 (10.8)

ADVERSE EVENTS:
Arm/Group | US-guided Group | Fluoroscopy-guided Group | Combined-guided Group
Serious Adverse Events (participants affected / at risk) | 0/147 | 0/145 | 0/146
Other Adverse Events (participants affected / at risk) | 17/147 | 31/145 | 20/146
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | US-guided Group (N=147) | Fluoroscopy-guided Group (N=145) | Combined-guided Group (N=146)
Perioperative complications (Surgical and medical procedures) | 17 | 31 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No